CLINICAL TRIAL: NCT02978911
Title: Diffusion Tensor Imaging and Tractography for Cranial Nerves. Interest in Skull Base Surgery and Anatomy
Brief Title: Cranial Nerves Tractography
Acronym: CN Tracto
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL16_0759; 2015-A01113-46 (Other: ID-RCB)
Record Dates: First submitted 2016-11-23; First posted 2016-12-01 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cranial Nerve Palsy
Keywords: RMI
MeSH Terms: conditions — Cranial Nerve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Skull base tumors (Experimental): Patients who presented a skull base tumor that requires a surgical removal
  Interventions: Procedure: preoperative cerebral MRI and operative findings

INTERVENTIONS:
Procedure: preoperative cerebral MRI and operative findings

SUMMARY:
Introduction: The skull base tumors surgery remains a challenge since numerous cranial nerves or vessels closely surround them. Recently, diffusion tensor imaging has developed with the tractography following white fibers and visualizing functional tracts. Cranial nerves tractography could allow predicting their displacement by skull base tumors that may help the surgeon to spare them along the surgery.

Methods: Preoperative cerebral MRI was performed on patients who presented with skull base tumors. A 3 tesla MRI machine was used to acquire DTI sequence with specific parameters: 32 directions, slice thickness 2 mm, echo time 86 ms, repetition time 12000 ms, matrix 128x128, b-value 1000 s.mm-1. An anatomic sequence hyperT2 was overlaid as reference. Distortion was corrected by topup and eddy functions from FSL. Cranial nerves fibers were probabilistically tracked with Mrtrix3. Cranial nerves were selected according to their location around the tumor. The "radiological" expected position of the cranial nerve was compared to its "operative" real position.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present a skull base tumor that requires surgical removal
* Patients adult, informed and agreed

Exclusion Criteria:

* Pregnant women
* Patients under 18 years old, unable to legally consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-07-12 (Actual); Primary Completion 2026-07-12 (Estimated); Study Completion 2026-07-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between the expected and the real position of the selected cranial nerve | Date of preoperative MRI (<3 months before the surgery)
  Selection of one or multiples cranial nerves of interest due to their close relationship with the tumor. Comparison of its/their position on MRI and during surgery.
Correlation between the expected and the real position of the selected cranial nerve | at 3 months
  Selection of one or multiples cranial nerves of interest due to their close relationship with the tumor. Comparison of its/their position on MRI and during surgery.

SECONDARY OUTCOMES:
postoperative cranial nerve palsy | at 3 months
  comparison with preoperative status

CONTACTS AND LOCATIONS:
Overall Officials: Timothée Jacquesson, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de Neurologie B, Hôpital Neurologique, HCL, Bron, France

IPD SHARING:
Plan to Share IPD: No